CLINICAL TRIAL: NCT02247245
Title: The Influence of Iatrogenic Chronotropic Incompetence on Exercise Tolerance in Pacemaker Patients With Chronic Heart Failure.
Brief Title: The Influence of Heart Rate Limitation on Exercise Tolerance in Pacemaker Patients.
Acronym: TREPPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Haqeel Jamil, Cardiology Registrar and Clinical Research Fellow, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LIGHT-TREPPE-1
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Chronic Heart Failure; Atrial Fibrillation; Arrhythmia, Sinus
Keywords: CHF; AF; SR; HFREF; CRT
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmia, Sinus | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects are given a placebo capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Interventions: Drug: Placebo
- Ivabradine (Active Comparator): Subjects are given an ivabradine capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Interventions: Drug: Ivabradine
- Atrial fibrillation (Experimental): Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algortithms switched on.
  Interventions: Other: Atrial fibrillation

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 7.5mg
  Other Names: Precorolan
  Arms: Ivabradine
Other: Atrial fibrillation — Pacemaker base rate alteration
  Arms: Atrial fibrillation
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To examine the effects of heart rate reduction on exercise capacity in control subjects and patients with chronic heart failure.

DETAILED DESCRIPTION:
Original proposal: Does iatrogenic chronotropic incompetence lead to impaired exercise capacity in patients with CHF

Aim The aim of this proposal is to examine the effects of iatrogenic CI on exercise capacity in control subjects and patients with chronic heart failure.

Hypothesis Iatrogenic chronotropic incompetence does not contribute significantly to reductions in exercise capacity in patients with heart failure or control subjects with pacemakers.

Methods REDUCING HEART RATE AT REST AND EXERCISE In patients with sinus rhythm, the present proposal utilizes a heart failure medication called ivabradine. This agent, an If channel blocker, specifically targets the sinus node leading to a slower heart rate. The agent is approved and licensed for use in patients with heart failure at the doses proposed. Ivabradine slows the sinus rate with none of the peripheral effects of beta-blockers. Heart rate lowering with ivabradine improves cardiac function, and outcomes related to the degree of bradycardia achieved.

In patients with atrial fibrillation, the present proposal will recruit patients with CRT and atrial fibrillation that have undergone atrio-ventricular node (AVN) ablation to improve the efficacy of CRT. Patients who have undergone AVN ablation are dependent upon their pacemaker, and we can therefore control their heart rate accurately.

SUBJECT SELECTION Inclusion criteria We will only include patients able to give informed written consent, which will be obtained in all subjects, and those capable of performing a peak exercise test. Since we are performing the study on three groups of patients, further inclusion criteria for each group are outlined below.

Inclusion criteria - CRT-sinus rhythm group We will enrol 25 patients with severe CHF on otherwise optimally tolerated medical therapy who have undergone cardiac resynchronisation therapy at least 3 months previously. These individuals will be on optimal medical therapy for their heart failure with no change in medication or exacerbation for the preceding 3 months. They will not currently be taking ivabradine.

Inclusion criteria - CRT-atrial fibrillation group We will enrol 25 patients with severe CHF on otherwise optimally tolerated medical therapy who have undergone cardiac resynchronisation therapy at least 3 months previously. All patients will be previously pacemaker dependant or have 'blocked' atrial fibrillation either due to medical therapy or previous atrio-ventricular nodal ablation.

Inclusion criteria - control group The control subjects (n=25) will be recruited from the general pacemaker clinic. They will undergo echocardiography to exclude structural heart disease. They will have no contraindications to exercise testing or ivabradine.

Exclusion criteria We will exclude subjects with musculoskeletal disorders limiting exercise capacity, patients with peripheral vascular disease, those with inflammatory disorders such as rheumatoid arthritis, and airways disease. Other exclusions include contraindications to ivabradine use such as severe hepatic impairment, significant renal impairment (creatinine clearance <15ml.min-1), and long QT syndrome. We will only include patients able to give informed written consent, which will be obtained in all subjects.

ECHOCARDIOGRAPHY Each subject will undergo a full echocardiographic examination. The images will be stored on a commercially available database, (Echopac PC, GE-Vingmed, USA) and analysed offline. We will assess LV systolic and diastolic function variables, mitral regurgitation, and pulmonary artery pressure.

EXERCISE TESTING Patients will describe their own NYHA symptom class at the beginning of each exercise session. Each individual will be invited for a familiarization test once agreeing to the study. At least one week following the familiarization test, heart failure patients and controls will return to the exercise laboratory and will be randomised to either ivabradine (7.5mg) or placebo. The following week they will return for the second arm. The randomization will be carried out in pharmacy to ensure blinding of the subject, the technician and the investigator. After ingesting the capsule, the subject will be asked to wait for an hour before the exercise test commences.

Prior to the start of exercise, patients' devices will be programmed to a base rate of 40 bts/min and they will then be they will be randomised to have their device programmed to either rate response on or off. A screen will separate the electrocardiographic monitor, which will be observed by the unblinded technician, from the metabolic cart, which will be observed by the blinded physician. The following week the other mode will be activated. At the end of each test the device will be returned to its original setting.

For the treadmill tests we will use the Bruce protocol modified by the addition of a 'stage 0' at onset consisting of 3 minutes of exercise at 1.61km/hr (1mile/hour) with a 5% gradient. During each test, expired air will be collected continuously and metabolic gas exchange analysis performed (Vmax 29, Sensormedics, USA). The system will be recalibrated prior to each test. Subjects will be encouraged to exercise to exhaustion, and a respiratory exchange ratio (RER), (VCO2/VO2) greater than 1.1 will be taken to suggest a maximal effort. The anaerobic threshold for each test will be calculated using the VO2/VCO2 slope method. At the end of each stage and at peak exercise subjects will be asked to indicate their score for dyspnoea or fatigue on a scale from 0 (no symptoms) to 10 (maximal symptoms) using the standardised Borg scoring system. The slope relating symptom scores against ventilation (Borg/VE) for each subject can then be plotted. We will also examine other ventilatory variables such as tidal volume (VT) and frequency (f) of ventilation.

ELIGIBILITY:
Inclusion criteria:

We will only include patients able to give informed written consent, which will be obtained in all subjects, and those capable of performing a peak exercise test. Since we are performing the study on three groups of patients, further inclusion criteria for each group are outlined below.

Inclusion criteria - CRT-sinus rhythm group We will enrol 25 patients with severe CHF on otherwise optimally tolerated medical therapy who have undergone cardiac resynchronisation therapy at least 3 months previously. These individuals will be on optimal medical therapy for their heart failure with no change in medication or exacerbation for the preceding 3 months. They will not currently be taking ivabradine.

Inclusion criteria - CRT-atrial fibrillation group We will enrol 25 patients with severe CHF on otherwise optimally tolerated medical therapy who have undergone cardiac resynchronisation therapy at least 3 months previously. All patients will be previously pacemaker dependant or have 'blocked' atrial fibrillation either due to medical therapy or previous atrio-ventricular nodal ablation.

Inclusion criteria - control group The control subjects (n=25) will be recruited from the general pacemaker clinic. They will undergo echocardiography to exclude structural heart disease. They will have no contraindications to exercise testing or ivabradine.

Exclusion Criteria:

We will exclude subjects with musculoskeletal disorders limiting exercise capacity, patients with peripheral vascular disease, those with inflammatory disorders such as rheumatoid arthritis, and airways disease. Other exclusions include contraindications to ivabradine use such as severe hepatic impairment, significant renal impairment (creatinine clearance <15ml.min-1), and long QT syndrome. We will only include patients able to give informed written consent, which will be obtained in all subjects.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus K Witte, FRCP MD, Principal Investigator — University of Leeds; Haqeel A Jamil, MbChB MRCP, Principal Investigator — University of Leeds
Locations (1):
- Leeds Institute of Cardiovascular and Metabolic Medicine, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Jamil HA, Gierula J, Paton MF, Byrom R, Lowry JE, Cubbon RM, Cairns DA, Kearney MT, Witte KK. Chronotropic Incompetence Does Not Limit Exercise Capacity in Chronic Heart Failure. J Am Coll Cardiol. 2016 Apr 26;67(16):1885-96. doi: 10.1016/j.jacc.2016.02.042. PMID 27102504

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The predicted group size to demonstrate a clinically important change was revised after post hoc analysis of pilot data demonstrating higher pVO2 values for both SR and AF than expected (minimum requirements:12 subjects in AF group, 20 in SR group). To allow for dropouts, recruitment targets were altered 14 with AF and 26 with SR (total 40).
Groups:
- Placebo First: Subjects are given a placebo capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Placebo: Placebo
  n=13 Placebo first, washout 1 week, then Ivabradine 7.5mg
- Ivabradine First: Subjects are given an ivabradine capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Ivabradine: Ivabradine 7.5mg
  Ivabradine 7.5mg first, washout 1 week, then placebo
- Atrial Fibrillation (Low Rate); Atrial Fibrillation (Standard Rate): Atrial fibrillation with pacemaker base rate alteration: Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algortithms switched on.
Period: Overall Study
Arm/Group | Placebo First | Ivabradine First | Atrial Fibrillation (Low Rate) | Atrial Fibrillation (Standard Rate)
Started | 13 | 13 | 7 | 7
Completed | 13 | 13 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo First: Subjects are given a placebo capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Placebo: Placebo
- Ivabradine First: Subjects are given an ivabradine capsule (double-blinded) to take 90 minutes prior to the cardiopulmonary exercise test.
  Ivabradine: Ivabradine 7.5mg
- Atrial Fibrillation (Low Rate): Atrial fibrillation with pacemaker base rate alteration: Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algortithms switched on.
  This group - low base pacing rate (30)
- Atrial Fibrilaltion (Standard Rate): Atrial fibrillation with pacemaker base rate alteration: Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algortithms switched on.
  This group - standard base pacing rate (60)
- Total: Total of all reporting groups
Arm/Group | Placebo First | Ivabradine First | Atrial Fibrillation (Low Rate) | Atrial Fibrilaltion (Standard Rate) | Total
Number analyzed (Participants) | 13 | 13 | 7 | 7 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (9) | 74 (9) | 76 (10) | 76 (10) | 74 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 2 | 10
  Male | 10 | 10 | 5 | 5 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 13 | 7 | 7 | 40
New York Heart Association classification [Median (Inter-Quartile Range); unit: units on a scale] — NYHA Stages of Heart Failure:
  Class 1 - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class 2 - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class 3 - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class 4 - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Higher class = worse outcomes
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Consumption (Peak VO2)
Description: Cardiopulmonary exercise testing performance - measuring peak oxygen uptake during a treadmill CPEX test.
  Subjects were exercised using the Bruce protocol, modified by the addition of a "stage 0" at onset consisting of 3 min of exercise at 1.61 km·h-1 (1 mile·h-1) with a 5% gradient. Expired air was collected and metabolic gas exchange analysis performed in order to measure the maximal oxygen consumption (peak VO2) (Sensormedics, Yorba Linda, California).
  The CPX equipment was recalibrated before every exercise test. All test subjects were encouraged to exercise to exhaustion before starting the test, and no further motivation or instructions were given.
Time Frame: Each test lasts up to 20 minutes
Measure: Mean (Standard Error); unit: ml/kg/min
Groups:
- Atrial Fibrillation: Low Base Rate (+no Rate Adaptive Pacing): Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algorithms switched on.
  Atrial fibrillation: Pacemaker base rate alteration
- Atrial Fibrn: Standard Base Rate (+Rate Adaptive Pacing): Subjects are (double blind) randomised to either a low base pacing rate (30) or a standard base rate (60), with rate adaptive algortithms switched on.
  Atrial fibrillation: Pacemaker base rate alteration
Arm/Group | Placebo | Ivabradine | Atrial Fibrillation: Low Base Rate (+no Rate Adaptive Pacing) | Atrial Fibrn: Standard Base Rate (+Rate Adaptive Pacing)
Number analyzed (Participants) | 13 | 13 | 7 | 7
ml/kg/min | 16 (3) | 17 (3) | 15.3 (1.9) | 14.2 (2.1)

ADVERSE EVENTS:
Time Frame: 2 weeks: immediate/early complications post intervention
Description: All-cause mortality, serious adverse events, non-serious/other adverse events
Groups:
- Atrial Fibrillation (Low Rate): Subjects are (double blind) randomised to a low base pacing rate (30) with rate adaptive algortithms switched on.
- Atrial Fibrilaltion (Standard Rate): Subjects are (double blind) randomised to a standard base pacing rate (60) with rate adaptive algortithms switched on.
Arm/Group | Placebo | Ivabradine | Atrial Fibrillation (Low Rate) | Atrial Fibrilaltion (Standard Rate)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes